CLINICAL TRIAL: NCT06986707
Title: Comparative Effects of Strain Counterstrain Technique and Graston Technique on Trigger Points of Quadratus Lumborum Among Patients With Nonspecific Low Back Pain
Brief Title: Strain Counterstrain Technique and Graston Technqiue on Quadratus Lumborum Trigger Points
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0157
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: low back pain; quadratus lumborum
MeSH Terms: conditions — Myofascial Pain Syndromes; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strain counterstrain technique (Experimental): Strain Counter-Strain Technique:
  (repeated 2 sets in each session)
  * 1 day per week
  * 4 weeks protocol
  Interventions: Other: Strain counterstrain technique
- Graston technique (Active Comparator): Before starting procedure, brisk walking or stretching is done for 4- 5 minutes
  * Applying heat for 3-4 minutes to warm the area
  * 40 seconds on right side
  * 40 seconds on left side
  Interventions: Other: Graston technique

INTERVENTIONS:
Other: Strain counterstrain technique — Group A: Conventional treatment will be given for 45 minutes (repeated 2 sets in each session)
  * 1 day per week
  * 4 weeks protocol
  Arms: strain counterstrain technique
Other: Graston technique — GROUP B: Conventional treatment will be given for 45 minutes Before starting procedure, brisk walking or stretching is done for 4- 5 minutes
  * Applying heat for 3-4 minutes to warm the area
  * 40 seconds on right side
  * 40 seconds on left side
  * 1 day per week
  * 4 weeks protocol After treatment, apply Ice for 2 minutes
  Arms: Graston technique

SUMMARY:
Poor body mechanics and posture affects body positioning and stresses quadratus lumborum muscle which ultimately leads to myofascial trigger points in muscle. This study aims to compare the effects of Strain counterstrain technique and Graston technique on trigger points of quadratus lumborum in nonspecific low back patients. This study will be a randomized controlled trial and will be conducted in Riphah Rehabilitation Clinic Lahore and SPARC Physiotherapy Clinic Lahore. Non-probability convenient sampling will be used to collect the data. Sample size of 34 subjects with age group between 20-45 years will be taken. baseline and after 4 weeks. Data analysis will be done by SPSS version 25.

DETAILED DESCRIPTION:
Researches have been conducted about effect of instrument assisted soft tissue mobilization versus kinesiotape for chronic mechanical low back pain: a randomized controlled trial. Introduction. The objective was to compare the effect of conventional program, instrument assisted soft tissue mobilization (IASTM) and kinesiotape (KT) in patients with chronic mechanical low back pain (CMLBP). 51 participants were randomly enrolled into three equal groups. Group A (n = 17) received conventional program, Group B (n = 17) received conventional program plus IASTM, and Group C (n = 17) received conventional program plus KT. The participants were evaluated before and after eight sessions using the Visual Analogue Scale (VAS), pressure algometer, dual inclinometer, and Oswestry Disability Index (ODI). It was concluded that Conventional program, IASTM and KT are effective methods for improving pain, ROM and function on CMLBP..Low back pain especially which is not related to any specific disease has become very common nowadays. Almost every other person complains about back pain. While there have been numerous studies on low back pain and its treatments but limited work has done on both techniques, the strain counterstrain technique and Graston technique. This study aims to determine the comparison of strain counterstrain technique and Graston technique on trigger points of quadratus lumborum among patients with non-specific low back pain

ELIGIBILITY:
Inclusion Criteria:

* Participant's age range 20-45 years
* Both genders.
* Individuals having low back pain for atleast 12 weeks with limited segmental mobility especially after maintaining certain prolonged posture .
* Individuals with localized pain and tenderness at attachments of quadratus lumborum due to the presence of trigger points (unilateral or bilateral).
* positive segmental mobility assessment at the level of L4 and L5 on one side or on both sides
* Patients having moderate pain on NPRS

Exclusion Criteria:

* Individuals with anticoagulation or bleeding disorders, acute muscle trauma, infections, lumbar disc herniation, spinal deformities, or a history of spinal surgery or anticoagulation medication
* Orthopedic surgery or any other low back surgery .
* Fracture of vertebrae and any lower limb injury

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | 4 weeks
  The Oswestry Disability Index (ODI) a patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. This is a 10-item index: 8 of them are related to activities of daily living and 2 refer to pain. The score of each item ranges from 0 to 5, with higher scores indicating greater disability. The total score is expressed as percentage

SECONDARY OUTCOMES:
Inclinometer | 4 weeks
  An inclinometer will be placed on the T12-L1 and L5-S1 spinal interspaces and zeroed with the patient in neutral standing position. The examiner asked the patient to bend forward maximally and then recorded the motion. Lumbar flexion will be represented by the difference in motion between the upper and lower inclinometers (12).
Numerical Pain Rating Scale (NPRS): | 4 weeks
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain"

CONTACTS AND LOCATIONS:
Overall Officials: Hira Shaukat, TDPT, Principal Investigator — Riphah International University
Locations (1):
- Kishwar sultana hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No